CLINICAL TRIAL: NCT07026188
Title: Clinical Evaluation of New Bone Formation During Limb Lengthening in Children by Ultrasound Combined With Superb Microvascular Imaging
Brief Title: Ultrasound Combined With SMI Imaging on Children With Limb Lengthening
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: ningbo1425
Record Dates: First submitted 2025-02-19; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Bone Anomalies
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bone-lengthening in children: Children who undergo bone-lengthening were taken US examination timely, to evaluate the bone recovering by one US doctor.
  Interventions: Other: Ultrasound with SMI

INTERVENTIONS:
Other: Ultrasound with SMI — The use of ultrasound allows observation of new bone formation in the distraction gap, also visualize the formation of blood vessels in the distraction gap with SMI, including the velocity and resistance of blood vessels, and can also indicate the environment of new bone formation. All US examination were performed by one US doctor.

SUMMARY:
In the present study, The use of ultrasound allows observation of new bone formation in the distraction gap, also visualize the formation of blood vessels in the distraction gap, including the velocity and resistance of blood vessels, and can also indicate the environment of new bone formation. It's considered that ultrasound detection of new bone and angiogenesis in the process of bone lengthening in children could be a good supplement to X-ray evaluation, and even partially replace the former, reducing the radiation burden of pediatric patients.

DETAILED DESCRIPTION:
Limb lengthening is one of most common surgical techniques for correcting limb deformities in pediatric patients. The evaluation of new bone formation in the distraction gap is very important for the prognosis of limb lengthening. After limb lengthening, weekly or biweekly plain X-ray is the most commonly-used method to evaluate new bone formation in the distraction gap. However, Ordinary X-ray (film or digital) cannot provide details of regeneration or vascular regeneration like ultrasound examination, and radiation damage caused by X-ray or CT has unpredictable negative effects on minors. Ultrasound and X-ray examination were performed every 2 weeks during lengthening in 30 pediatric patients. Ultrasound was used to observe the formation of new bone, the number of vertical vessels and the blood flow resistance index, which were compared with the corresponding X-ray findings.New bone states could be divided by US into three stages: stage I (early lengthening): no obvious callus formation was found X-ray and ultrasound; stage II (lengthening stage): X-ray showed low density callus formation and uneven density, which was divided into three stages by ultrasound: IIa, punctate callus could be seen; IIb, linear callus was found, but not connected; IIc, connected linear callus was found; stage III (healing stage): the broken ends of the bone were joined, the periosteum was continuous, and the callus had disappeared. X-ray showed healing of the lengthened bone.

ELIGIBILITY:
Inclusion Criteria:

* All are children who suffer limb length discrepancy and need limb-lengthening procedure; with no difference in sex, age or ethics.

Exclusion Criteria:

* Space of braces is smaller than the probes.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All are children who suffer limb length discrepancy and need limb-lengthening procedure; with no difference in sex, age or ethics.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Gray scale of US in bone gap. | From the first day of lengthening to the removal of the external fixator.（Approximately 6 months.）
  New bone states were divided into three stages: stage I (early lengthening): no obvious callus formation was found X-ray and ultrasound; stage II (lengthening stage): X-ray showed low density callus formation and uneven density, which was divided into three stages by ultrasound: IIa, punctate callus could be seen; IIb, linear callus was found, but not connected; IIc, connected linear callus was found; stage III (healing stage): the broken ends of the bone were joined, the periosteum was continuous, and the callus had disappeared.
New vessels of bone gap. | From the first day of lengthening to the removal of the external fixator.（Approximately 6 months.）
  The number of vessels in the lengthening gap, assessed via ultrasound techniques like SMI, reflects the vertical vessels growing into the distraction gap. This metric offers insights into the microvascular environment and angiogenesis of the new bone, aiding in evaluating healing progress and guiding lengthening protocol adjustments.
Resistance index of new vessles. | From the first day of lengthening to the removal of the external fixator.（Approximately 6 months.）
  The resistance index of new vessels, measured using ultrasound techniques like SMI, assesses blood flow resistance in the newly formed vessels within the lengthening gap.
Healing index | From the first day of lengthening to 2 months after the removal of the external fixator.（Approximately 8 months.）
  The healing index, calculated as healing time in months divided by lengthening distance in centimeters, serves as an objective indicator of limb lengthening prognosis. A smaller healing index signifies a faster healing rate.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Bo, MD, Principal Investigator — Pediatric hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No